CLINICAL TRIAL: NCT04160078
Title: Adapting a Mindfulness Intervention to Improve Sleep and Reduce Diabetes Risk Among a Diverse Sample in Atlanta
Brief Title: Mindfulness IN-home for Diabetes and Sleep Health
Acronym: MINDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Center for Diabetes Translation Research (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Dayna A. Johnson, Assistant professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00112861; P30DK111024 (NIH)
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
Keywords: Diabetes; Mindfulness; Public health; Sleep
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Mindfulness-Based Stress Reduction; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Intervention Arm (Experimental): A stress reduction plus sleep education intervention to improve sleep health
  Interventions: Behavioral: Mindfulness-based stress reduction (MBSR) Intervention

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction (MBSR) Intervention — * 1-hour session on sleep hygiene and 7-week follow up using a mindfulness app, an app that features guided meditation and can be used to assess adherence.
  * Sleep log diary: self report of sleep records
  * Wrist Actigraphy, to monitor sleep patterns. Participants will be instructed on wearing the sleep monitor (Spectrum, Philips Respironics, Murrysville, PA) on their non-dominant wrist for the next 7-weeks
  Other Names: MBSR Intervention

SUMMARY:
The study investigates the effects of a mindfulness intervention on sleep and subsequent cardio-metabolic risk in an adult Atlanta population aged 18 and older.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus has been identified as a leading cause of death in the United States. This problem is alarmingly higher in southern state, including Georgia. Sleep, a modifiable health behavior, may be a target for reducing the burden of diabetes. This research study will enroll adults from the community to participate in a mindfulness-based stress reduction program (MBSR) via an app on his/her cellular phone. Participants will also wear a wrist monitor to estimate activity and sleep as well as provide a blood sample before and after the MBSR. Following the 6-week intervention program, participants will provide information via focus groups to obtain feedback on his/her experiences during the program.

This pilot study will enroll (N=20) racially diverse men and women who are 18 years and older and reside in Atlanta. Participants will be recruited from the community via advertisements, community events and existing community partnerships. Trained research assistants will screen potential participants. Eligible participants will be contacted via phone and scheduled to attend a baseline visit to collect a blood sample and attend a sleep education session.

ELIGIBILITY:
Inclusion Criteria:

* Resident in the Atlanta, Georgia area
* Proficient in English
* Have a smartphone
* Sleep quality score >5 on the validated Pittsburgh Sleep Quality Index
* Prediabetes (defined as fasting glucose between 100-125 mg/dL or HbA1c between 5.7-6.4%)

Exclusion Criteria:

* Pregnant women
* Sleep quality score less than a score 5 on the validated Pittsburgh Sleep Quality Index
* Refusal to download Mindfulness mobile application
* Diagnosis of HIV, AIDS, Liver disease (diagnosed, i.e. chronic or alcoholic hepatitis, cirrhosis), Renal/Kidney disease
* Current Cocaine, heroin, or methamphetamines use and/or has a history of treatment for alcohol or drug abuse
* Pre-diabetes: defined as a score greater than 3 on the American Diabetes Association 60-Second Type 2 Diabetes Risk Test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dayna Johnson, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Statistical analysis plan will be available upon request. Data will be available one year after the first person is enrolled with no end date.
Supporting Information: SAP
Time Frame: One year after the first person is enrolled. No end date.
Access Criteria: Researchers upon request will be able to access data, for any purpose. Data will be shared via secure data transfer.

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindfulness-based Stress Reduction (MBSR) Intervention: Participants receiving a stress reduction plus sleep education intervention to improve sleep health
Period: Overall Study
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.89 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2
  Race: Black or African American | 8
  Race: White | 6
  Race: Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
Education [Count of Participants; unit: Participants]
  Less than Bachelor's degree | 2
  Bachelor's degree | 9
  Professional degree (Master's, MD, PhD, law degree) | 7

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index (PSQI) Score
Description: Global sleep quality was measured via the validated Pittsburgh Sleep Quality Index (PSQI). The PSQI is a self-rated questionnaire which assesses several dimensions of sleep including sleep quality, duration, and disturbances over a 1-month time interval. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score which ranges from 0 to 21. Poor sleep quality is defined as a global score of 5 or greater.
Time Frame: Baseline, 4 weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
Number analyzed (Participants) | 18
score on a scale
  Baseline | 7.22 (2.96)
  4 weeks post-intervention | 5.00 (2.20)

2. Primary Outcome: Sleep Duration
Description: Sleep duration was measured in hours and minutes using a sleep 7-day actigraphy (Philips Respironics Actiwatch Spectrum Plus) on the non-dominant wrist, and confirmed with daily sleep logs. Self-reported sleep duration was also measured.
Time Frame: Baseline, 4 weeks post-intervention
Population: Some participants did not complete the 7-day actigraphy assessment.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
Number analyzed (Participants) | 18
hours
  Baseline assessed by actigraphy: number analyzed (Participants) | 17
  Baseline assessed by actigraphy | 6.19 (1.05)
  4 weeks post-intervention assessed by actigraphy: number analyzed (Participants) | 16
  4 weeks post-intervention assessed by actigraphy | 6.18 (1.45)
  Baseline assessed by self-report | 8.30 (1.33)
  4 weeks post-intervention assessed by self-report | 8.15 (1.82)

3. Primary Outcome: Perceived Stress Scale (PSS)
Description: The perceived stress scale is a validated tool to help understand how different situations affect feelings and perceived stress. The PSS has 10 items which are responded to on a 5-point scale where 0 = never and 4 = very often. Total scores range from 0 to 40 and higher scores indicate higher perceived stress.
Time Frame: Baseline, 4 weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
Number analyzed (Participants) | 18
score on a scale
  Baseline | 15.72 (7.73)
  4 weeks post-intervention | 13.44 (7.47)

4. Primary Outcome: Number of Participants With PSS Score Indicating Low Stress
Description: The perceived stress scale is a validated tool to help understand how different situations affect feelings and perceived stress. The PSS has 10 items which are responded to on a 5-point scale where 0 = never and 4 = very often. Total scores range from 0 to 40 and higher scores indicate higher perceived stress. Participants with scores of 0 to 13 are categorized as having low stress.
Time Frame: Baseline, 4 weeks post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
Number analyzed (Participants) | 18
Participants
  Low stress at Baseline | 7
  Low stress at 4 weeks post-intervention | 10

5. Primary Outcome: Number of Participants With PSS Score Indicating Moderate Stress
Description: The perceived stress scale is a validated tool to help understand how different situations affect feelings and perceived stress. The PSS has 10 items which are responded to on a 5-point scale where 0 = never and 4 = very often. Total scores range from 0 to 40 and higher scores indicate higher perceived stress. Participants with scores of 14 to 26 are categorized as having moderate stress.
Time Frame: Baseline, 4 weeks post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
Number analyzed (Participants) | 18
Participants
  Moderate stress at Baseline | 10
  Moderate stress at 4 weeks post-intervention | 8

6. Primary Outcome: Number of Participants With PSS Score Indicating High Stress
Description: The perceived stress scale is a validated tool to help understand how different situations affect feelings and perceived stress. The PSS has 10 items which are responded to on a 5-point scale where 0 = never and 4 = very often. Total scores range from 0 to 40 and higher scores indicate higher perceived stress. Participants with scores of 27 to 40 are categorized as having high stress.
Time Frame: Baseline, 4 weeks post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
Number analyzed (Participants) | 18
Participants
  High stress at Baseline | 1
  High stress at 4 weeks post-intervention | 0

7. Secondary Outcome: Weight
Description: Participants provided their weight in pounds (lbs) based on a scale that was distributed to participants.
Time Frame: Baseline, 4 weeks post-intervention
Population: One participant did not report weight at the 4 week post-intervention assessment.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
Number analyzed (Participants) | 18
pounds
  Baseline | 180.64 (30.00)
  4 weeks post-intervention: number analyzed (Participants) | 17
  4 weeks post-intervention | 184.12 (29.77)

8. Secondary Outcome: Body Mass Index (BMI)
Description: Body mass index (BMI) is calculated as weight in kilograms (kg) divided by the square of the body height measured in meters (m). A BMI between 18.5 and 24.9 is considered to be normal weight. A BMI of 25-29.9 indicates overweight, while a BMI of 30 or more indicates obesity.
Time Frame: Baseline, 4 weeks post-intervention
Population: One participant did not report weight at the 4 weeks post-intervention assessment.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
Number analyzed (Participants) | 18
kg/m^2
  Baseline | 29.93 (5.22)
  4 weeks post-assessment | 30.21 (5.27)

9. Secondary Outcome: Blood Pressure
Description: Blood pressure is the pressure of circulating blood on the walls of blood vessels and is measured in millimeters of mercury (mmHg). Three seated blood pressure measurements were made using an electronic sphygmomanometer. An average of the last two readings were used to assess systolic and diastolic blood pressure. Blood pressure values of less than 120 mmHg systolic and 80 mmHg diastolic are considered within the normal range.
Time Frame: Baseline, 4 weeks post-intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
Number analyzed (Participants) | 18
mmHg
  Systolic blood pressure at Baseline | 110.03 (11.13)
  Systolic blood pressure at 4 weeks post-intervention | 112.47 (8.90)
  Diastolic blood pressure at Baseline | 70.31 (8.14)
  Diastolic blood pressure at 4 weeks post-intervention | 71.06 (6.99)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time of participant consent through the follow up visit at 4 weeks post-intervention.
Arm/Group | Mindfulness-based Stress Reduction (MBSR) Intervention
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mindfulness-based Stress Reduction (MBSR) Intervention (N=18)
Rash from sleep monitor wrist band (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT04160078/Prot_SAP_001.pdf
  • Informed Consent Form (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT04160078/ICF_000.pdf